CLINICAL TRIAL: NCT03147326
Title: The Diagnostic Value of FDG-PET-CT, NaF-PET-CT and Whole-body MRI Compared to Whole-body Xray in the Detection of Bone Lesions in Multiple Myeloma Patients
Brief Title: Diagnostic Imaging of Myeloma Bone Lesions
Acronym: RAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Eva Dyrberg Mortensen, Medical doctor, PhD-student, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAMP
Record Dates: First submitted 2017-04-25; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG-NaF-MRI (Other): All participants will undergo three project scans/the following interventions:
  FDG-PET-CT NaF-PET-CT Whole-body MRI All participants will undergo a whole-body x-ray as part of clinical routine practice.
  Interventions: Diagnostic Test: FDG-PET-CT; Diagnostic Test: NaF-PET-CT; Diagnostic Test: Whole-body MRI

INTERVENTIONS:
Diagnostic Test: FDG-PET-CT — scanning method
Diagnostic Test: NaF-PET-CT — scanning method
Diagnostic Test: Whole-body MRI — scanning method

SUMMARY:
The purpose of this study is to compare the current standard whole-body x-ray with the advanced imaging techniques FDG-PET-CT, NaF-PET-CT and whole-body MRI in the detection of myeloma bone lesions.

DETAILED DESCRIPTION:
Accurate detection of bone lesions in myeloma patients is essential for treatment planning and patient survival.

Newly diagnosed multiple myeloma patients can be enrolled in this study. All participants will at time of diagnosis undergo three project scans (FDG-PET-CT, NaF-PET-CT, whole-body MRI) as well as whole-body x-ray as part of clinical routine practice.

Experienced specialists in the field of radiology and nuclear medicine interpret the images. Each reader performs the evaluations blinded to other imaging results as well as to the patient's clinical information. The reader assesses whether myeloma indicative bone lesions are present in eight predefined skeletal body regions.

Endpoint is purely diagnostic.

Statistics:

Cochran's Q-test: to compare the proportion of patients with bone disease detected by the four scanning methods.

Two-sided ANOVA: to compare the average number of regions detected with bone disease by the four scanning methods.

Tukey's comparison test: to compare the difference between each pair of means.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma (biopsy proven)

Exclusion Criteria:

* Prior malignancy
* Are not able to undergo a MRI scan due to MRI contraindications (e.g. pacemaker)
* Has any condition that places the subject at an unacceptable risk if he/she undergoes a diagnostic CT scan with iv. contrast (e.g. history of severe allergic reaction to the contrast agent)
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Bone metastases detection rate - a patient-based analysis | The three project scans will be performed once and as baseline scans within a maximum of 30 days from the performance of the whole-body x-ray. Image analyses and statistical tests will be done when all project scans have been performed
  To compare the proportion of patients with bone disease detected by the four scanning techniques
Bone metastases detection rate - a region-based analysis | The three project scans will be performed once and as baseline scans within a maximum of 30 days from the performance of the whole-body x-ray. Image analyses and statistical tests will be done when all project scans have been performed
  To compare the number of affected regions with bone disease detected by the four scanning techniques

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S. Thomsen, Professor, Study Director — Department of Radiology
Locations (1):
- Department of Radiology/Department of Nuclear Medicine, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No